CLINICAL TRIAL: NCT01270022
Title: Development, Implementation and Evaluation of the Impact of a Guideline in Clinical Practise for Cardiovascular Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia De Atencion Primaria Area 2 De Madrid (Other Government)
Collaborators: Health Research Fund of ISCIII Spain (Unknown)
Responsible Party: Blanca Novella Arribas, Gerencia de Atención Primaria Area 2 Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PI031216
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Cardiovascular Risk Factors; Clinical Practice Guideline; Implementation Strategies; Primary Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Implementation (Experimental)
  Interventions: Other: Implementation
- dissemination (Active Comparator)
  Interventions: Other: dissemination

INTERVENTIONS:
Other: Implementation
  Arms: Implementation
Other: dissemination
  Arms: dissemination

SUMMARY:
The aim of this study is to evaluate the impact of a clinical guideline in cardiovascular risk, with a local adaptation model of the existing guidelines in clinical practise at present, of each of the different cardiovascular risk factors, and the implementation strategy.

DETAILED DESCRIPTION:
With this objective this study will be developed in three diferent phases. The guideline in clinical practice elaboration. It will be based in evidence medicine and it will be adapted based in the cardiovascular risk factors guidelines published at the present.

The spreding and implementation of the guideline between the sanitarians, as much in primary medicine as in specialised area, involved in the care of the patient in cardiovascular risk, in the Area 2 in Madrid.

And the evaluation of the implementation strategy, used between the primary care physicians.

For the local adaptation, will be used a systematic review of the different guidelines in the Spanish and international literature, published in the last years about this topic.

The ones with better quality criteria will be selected and doctors and nurses related from different specialities, involved in the cardiovascular illness, as much as members of the staff of the medical management an nursery, will be invited to participate in the selection of the recommendations of the guides and in the search of the consensus. After that, this guide will be given to a group of patients, who will be asked for a critical approach and their suggestions will be applied.

The evaluation will be done with a clinical trial designe , testing the use of the guide and its results on health intermediary variables. With this objective the results with an implementation technique based on opinion leaders plus computer reminder, will be evaluated, instead of using the standard implementation.

ELIGIBILITY:
Inclusion Criteria:

* patients whose health cards showed them to belong to the studied health area

Exclusion Criteria:

* Clinical history have not opened in the health center or this one is empty

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Novella, MD. pHD, Principal Investigator — Gerencia de Atención Primaria del área 2
Locations (1):
- Gerencia de Atención Primaria del área 2, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Rodriguez-Salvanes F, Novella B, Fernandez Luque MJ, Sanchez-Gomez LM, Ruiz-Diaz L, Sanchez-Alcalde R, Sierra-Garcia B, Mayayo S, Ruiz-Lopez M, Loeches P, Lopez-Gonzalez J, Gonzalez-Gamarra A; SIRVA2 group. Efficacy of a strategy for implementing a guideline for the control of cardiovascular risk in a primary healthcare setting: the SIRVA2 study a controlled, blinded community intervention trial randomised by clusters. BMC Fam Pract. 2011 Apr 19;12:21. doi: 10.1186/1471-2296-12-21. PMID 21504570